CLINICAL TRIAL: NCT05576766
Title: Impact of Enhanced Recovery After Surgery (ERAS) Pathway on Outcomes in Patients Undergoing Robot-Assisted Laparoscopic Radical Prostatectomy: A Randomized Controlled Trial
Brief Title: Enhanced Recovery After Surgery (ERAS) Pathway in Patients Undergoing Robot-Assisted Laparoscopic Radical Prostatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-235
Record Dates: First submitted 2022-09-12; First posted 2022-10-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Robot-Assisted Laparoscopic Radical Prostatectomy; Enhanced Recovery After Surgery (ERAS) Protocol; Prehabilitation; Length of Hospital Stay
Keywords: Prostate Cancer; Robot-Assisted Laparoscopic Radical Prostatectomy; RARP; Enhanced Recovery After Surgery; ERAS; Prehabilitation; Length of hospital stay
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine care group (Active Comparator): Perioperative management according to routine care.
  Interventions: Procedure: Routine care
- ERAS group (Experimental): Perioperative management according to the Enhanced Recovery after Surgery (ERAS) pathway.
  Interventions: Procedure: ERAS management pathway

INTERVENTIONS:
Procedure: Routine care — 1. Routine information provided before surgery.
  2. No nutritional therapy.
  3. No aerobic exercise.
  4. No pelvic floor muscle training.
  5. No psychiatrist intervention.
  6. Bowel preparation with oral cathartic agent.
  7. Fasting for over 8 hours; no oral carbohydrate solution (OCS) loading before surgery.
  8. Hypothermia prevention not emphasized.
  9. General anesthesia; regional block not emphasized.
  10. Routine blood pressure management.
  11. Mobilization from postoperative day 1.
  12. Start oral feeding from postoperative day 1.
  13. Patient-controlled analgesia with opioids.
  14. Thromboembolism prophylaxis with low-molecular-weight heparin (LMWH).
  15. Routine pelvic drainage tube removal (usually at postoperative day 4).
  16. Routine urinary catheterization removal (usually at postoperative day 14).
  Arms: Routine care group
Procedure: ERAS management pathway — 1. Patient consultation and education before surgery.
  2. Nutritional intervention for patients whose BMI<18.5 or BMI>24 kg/m2.
  3. Aerobic exercise for 2 weeks before surgery.
  4. Pelvic floor muscle training for 2 weeks before surgery.
  5. Psychiatrist intervention for patients with severe depression and anxiety.
  6. No bowel preparation before surgery.
  7. Provide oral carbohydrate solution 2 hours before surgery.
  8. Hypothermia prevention.
  9. General anesthesia combined with regional block.
  10. Goal-directed fluid infusion and targeted blood pressure management.
  11. Early mobilization.
  12. Early oral feeding.
  13. Multimodal analgesia, including opioids and non-steroid anti-inflammatory drugs.
  14. Thromboembolism prophylaxis with low-molecular-weight heparin; rivaroxaban for high-risk patients.
  15. Early pelvic drainage tube removal (at postoperative day 2) unless contraindicated.
  16. Early urinary catheterization removal (at postoperative day 7) unless contraindicated.
  Arms: ERAS group

SUMMARY:
Prostate cancer ranks second among all malignances in men and has become a significant threat to men's health. Robot-assisted laparoscopic radical prostatectomy (RARP) has become a standard treatment for prostate cancer. How to improve recovery following RARP surgery is worth investigating. The enhanced recovery after surgery (ERAS) pathway involves a series of evidence-based procedures. It is aimed to reduce the systemic stress response to surgery and shorten the length of hospital stay. This randomized trial aims to investigate the impact of Enhanced Recovery After Surgery (ERAS) Pathway on early outcomes after RARP surgery.

DETAILED DESCRIPTION:
Prostate cancer ranks second among all malignancies in men and has become a significant threat to men's health. Surgical resection is the main treatment for patients with early and locally advanced prostate cancer. With the progress of technology, robot-assisted laparoscopic radical prostatectomy (RARP) is gradually accepted by surgeons and become the first line treatment for prostate cancer. How to improve recovery after RARP surgery is worth investigating.

The concept of enhanced recovery after surgery (ERAS) was first reported by Dr. Kehlet. The ERAS pathway involves a series of evidence-based managements to accelerate patients' rehabilitation, including selective bowel preparation, nutritional therapy, fluid management, multimodal analgesia, early mobilization, etc. It has been applied to many patient populations including those undergoing gastrointestinal surgery, cardiothoracic surgery, and urological surgery. Previous studies showed that practicing ERAS in patients undergoing laparoscopic prostate surgery shortened the time to flatus and defecate and the length of hospital stay. Specifically, prehabilitation including aerobic exercise and pelvic floor training may be beneficial and improve physical wellbeing in patients undergoing prostatectomy. However, little is known regarding the effects of ERAS in patients undergoing RARP surgery.

The purpose of this randomized controlled trial is to investigate the impact of ERAS management, including prehabilitation, on early outcomes in patients undergoing RARP surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or over but below 90 years.
* Scheduled to undergo robot-assisted laparoscopic radical prostatectomy (RARP) for prostate cancer.
* Agree to participate in this study and give written informed consent.

Exclusion Criteria:

* Scheduled to undergo combined surgery, including RARP combined with pelvic lymph node dissection or other procedures.
* American Society of Anesthesiologists (ASA) physical classification ≥IV.
* Inability to receive preoperative aerobic exercise because of severe cardiovascular disease, motor system diseases (arthritis, lumbar vertebrae disease), or central nervous system diseases (epilepsy, parkinsonism).
* Inability to communicate in the preoperative period because of profound dementia, deafness, or language barriers.
* History of schizophrenia, anxiety or depressive disorders, or other mental disorders.

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The time required for the PADS score to meet the standard. | Up to 30 days after surgery.
  The time required to achieve a post-anesthesia discharge score (PADS) of 9 or above after surgery.

SECONDARY OUTCOMES:
Perioperative anxiety score | On the day before surgery and at day 1 after surgery.
  The score of anxiety is assessed by using the Self-Rating Anxiety Scale (SAS). This is a 20-item self-report questionnaire; each item is rated from 1 to 4 denoting the increasing severity or frequency of anxiety; the sum score times 1.25 as a standard score, ranging from 25 to 100, with higher score indicating more severe anxiety.
Perioperative depression score | On the day before surgery and at day 1 after surgery.
  The score of depression is assessed by using the Self-Rating Depression Scale (SDS). This is a 20-item self-report questionnaire; each item is rated from 1 to 4 denoting the increasing severity or frequency of depression; the sum score times 1.25 as a standard score, ranging from 25 to 100, with higher score indicating more severe depression.
Pain score within 3 days after surgery | Up to 3 days after surgery
  Pain score is assessed twice daily (8:00-10:00 am, and 18:00-20:00 pm) with the Numeric Rating Scale (NRS), an 11-point scale ranging from 0 to 10, with 0=no pain and 10=the worst pain.
Incidence of postoperative complications within 30 days after surgery | Up to 30 days after surgery
  Postoperative complications are defined as new-onset medical events that are harmful to patients' recovery and required therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
Incidence of readmission within 30 days after surgery | Up to 30 days after surgery
  Readmission is defined as hospitalization for the second time after discharge within 30 days after surgery.
Overall survival within 90 days after surgery | Up to 90 days after surgery
  Overall survival within 90 days after surgery.
Total hospitalization cost within 30 days after surgery | Up to 30 days after surgery
  Total hospitalization cost is defined as the sum cost of hospitalization from admission up to 30 days after surgery, including re-hospitalization within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott JM, Zabor EC, Schwitzer E, Koelwyn GJ, Adams SC, Nilsen TS, Moskowitz CS, Matsoukas K, Iyengar NM, Dang CT, Jones LW. Efficacy of Exercise Therapy on Cardiorespiratory Fitness in Patients With Cancer: A Systematic Review and Meta-Analysis. J Clin Oncol. 2018 Aug 1;36(22):2297-2305. doi: 10.1200/JCO.2017.77.5809. Epub 2018 Jun 12. PMID 29894274
- [Background] Xing J, Wang J, Liu G, Jia Y. Effects of enhanced recovery after surgery on robotic radical prostatectomy: a systematic review and meta-analysis. Gland Surg. 2021 Dec;10(12):3264-3271. doi: 10.21037/gs-21-699. PMID 35070886
- [Background] Xu Y, Liu A, Chen L, Huang H, Gao Y, Zhang C, Xu Y, Huang D, Xu D, Zhang M. Enhanced recovery after surgery (ERAS) pathway optimizes outcomes and costs for minimally invasive radical prostatectomy. J Int Med Res. 2020 Jun;48(6):300060520920072. doi: 10.1177/0300060520920072. PMID 32485118
- [Background] Sugi M, Matsuda T, Yoshida T, Taniguchi H, Mishima T, Yanishi M, Komai Y, Yasuda K, Kinoshita H, Yoshida K, Watanabe M. Introduction of an Enhanced Recovery after Surgery Protocol for Robot-Assisted Laparoscopic Radical Prostatectomy. Urol Int. 2017;99(2):194-200. doi: 10.1159/000457805. Epub 2017 Feb 17. PMID 28222423
- [Background] Visioni A, Shah R, Gabriel E, Attwood K, Kukar M, Nurkin S. Enhanced Recovery After Surgery for Noncolorectal Surgery?: A Systematic Review and Meta-analysis of Major Abdominal Surgery. Ann Surg. 2018 Jan;267(1):57-65. doi: 10.1097/SLA.0000000000002267. PMID 28437313
- [Background] Kehlet H, Mogensen T. Hospital stay of 2 days after open sigmoidectomy with a multimodal rehabilitation programme. Br J Surg. 1999 Feb;86(2):227-30. doi: 10.1046/j.1365-2168.1999.01023.x. PMID 10100792
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Magheli A, Knoll N, Lein M, Hinz S, Kempkensteffen C, Gralla O. Impact of fast-track postoperative care on intestinal function, pain, and length of hospital stay after laparoscopic radical prostatectomy. J Endourol. 2011 Jul;25(7):1143-7. doi: 10.1089/end.2011.0020. PMID 21740262
- [Background] Lv Z, Cai Y, Jiang H, Yang C, Tang C, Xu H, Li Z, Fan B, Li Y. Impact of enhanced recovery after surgery or fast track surgery pathways in minimally invasive radical prostatectomy: a systematic review and meta-analysis. Transl Androl Urol. 2020 Jun;9(3):1037-1052. doi: 10.21037/tau-19-884. PMID 32676388
- [Background] Lin C, Wan F, Lu Y, Li G, Yu L, Wang M. Enhanced recovery after surgery protocol for prostate cancer patients undergoing laparoscopic radical prostatectomy. J Int Med Res. 2019 Jan;47(1):114-121. doi: 10.1177/0300060518796758. Epub 2018 Sep 9. PMID 30198392
- [Background] Milliken D, Lawrence H, Brown M, Cahill D, Newhall D, Barker D, Ayyash R, Kasivisvanathan R. Anaesthetic management for robotic-assisted laparoscopic prostatectomy: the first UK national survey of current practice. J Robot Surg. 2021 Jun;15(3):335-341. doi: 10.1007/s11701-020-01105-3. Epub 2020 Jun 24. PMID 32583048
- [Background] Santa Mina D, Hilton WJ, Matthew AG, Awasthi R, Bousquet-Dion G, Alibhai SMH, Au D, Fleshner NE, Finelli A, Clarke H, Aprikian A, Tanguay S, Carli F. Prehabilitation for radical prostatectomy: A multicentre randomized controlled trial. Surg Oncol. 2018 Jun;27(2):289-298. doi: 10.1016/j.suronc.2018.05.010. Epub 2018 May 7. PMID 29937184
- [Background] Zhao Y, Zhang S, Liu B, Li J, Hong H. Clinical efficacy of enhanced recovery after surgery (ERAS) program in patients undergoing radical prostatectomy: a systematic review and meta-analysis. World J Surg Oncol. 2020 Jun 17;18(1):131. doi: 10.1186/s12957-020-01897-6. PMID 32552894
- [Background] Segal RJ, Reid RD, Courneya KS, Sigal RJ, Kenny GP, Prud'Homme DG, Malone SC, Wells GA, Scott CG, Slovinec D'Angelo ME. Randomized controlled trial of resistance or aerobic exercise in men receiving radiation therapy for prostate cancer. J Clin Oncol. 2009 Jan 20;27(3):344-51. doi: 10.1200/JCO.2007.15.4963. Epub 2008 Dec 8. PMID 19064985
- [Background] Angenete E, Angeras U, Borjesson M, Ekelund J, Gellerstedt M, Thorsteinsdottir T, Steineck G, Haglind E. Physical activity before radical prostatectomy reduces sick leave after surgery - results from a prospective, non-randomized controlled clinical trial (LAPPRO). BMC Urol. 2016 Aug 16;16(1):50. doi: 10.1186/s12894-016-0168-0. PMID 27531014
- [Background] Liu Z, Qiu T, Pei L, Zhang Y, Xu L, Cui Y, Liang N, Li S, Chen W, Huang Y. Two-Week Multimodal Prehabilitation Program Improves Perioperative Functional Capability in Patients Undergoing Thoracoscopic Lobectomy for Lung Cancer: A Randomized Controlled Trial. Anesth Analg. 2020 Sep;131(3):840-849. doi: 10.1213/ANE.0000000000004342. PMID 31348053
- [Background] Hori T, Makino T, Fujimura R, Takimoto A, Urata S, Miyagi T. Favorable Impact on Postoperative Abdominal Symptoms in Robot-assisted Radical Prostatectomy Using Enhanced Recovery After Surgery Protocol. Cancer Diagn Progn. 2022 Mar 3;2(2):247-252. doi: 10.21873/cdp.10101. eCollection 2022 Mar-Apr. PMID 35399176
- [Background] Cao J, Gu J, Wang Y, Guo X, Gao X, Lu X. Clinical efficacy of an enhanced recovery after surgery protocol in patients undergoing robotic-assisted laparoscopic prostatectomy. J Int Med Res. 2021 Aug;49(8):3000605211033173. doi: 10.1177/03000605211033173. PMID 34423666